CLINICAL TRIAL: NCT00293319
Title: I-Metaiodobenzylguanidine (I-MIBG) Therapy for Refractory Neuroblastoma, A Phase II Study
Brief Title: 131 I-MIBG in Treating Patients With Refractory or Relapsed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine Matthay, Professor, Department of Pediatrics, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454716; UCSF-05161; UCSF-00161
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; 3-Iodobenzylguanidine

INTERVENTIONS:
Biological: filgrastim
Radiation: iobenguane I 131

SUMMARY:
RATIONALE: Radioactive drugs, such as 131 I-MIBG, may carry radiation directly to tumor cells and not harm normal cells.

PURPOSE: This phase II trial is studying how well 131 I-MIBG works in treating patients with refractory or relapsed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if iodine I 131 metaiodobenzylguanidine can provide palliative therapy for patients with refractory or relapsed neuroblastoma.
* Determine the acute and late toxicity of this regimen in these patients.

Secondary

* Determine disease and symptom responses of patients treated with this regimen.

OUTLINE: This is a compassionate use study.

Patients receive iodine I 131 metaiodobenzylguanidine IV over 2 hours. Beginning 10 days later, patients with low neutrophil counts receive filgrastim (G-CSF) subcutaneously until blood count recovers. Patients with stable or responding disease may receive a second dose of iodine I 131 metaiodobenzylguanidine at least 6 weeks after the first dose.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Original diagnosis of neuroblastoma based on 1 of the following criteria:

  * Histopathology
  * Elevated urine catecholamines with typical tumor cells in the bone marrow
* Refractory or relapsed disease, meeting 1 of the following criteria:

  * Failure to respond to standard therapy (e.g., combination chemotherapy with or without radiotherapy and surgery)
  * Evidence of disease progression (i.e., any new lesion or an increase in size of > 25% of a pre-existing lesion) at any time
* Evaluable disease by MIBG scan within 6 weeks of study entry

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* Bilirubin < 2 times normal
* AST/ALT ≤ 10 times normal
* Creatinine ≤ 2 mg/dL
* Absolute neutrophil count* ≥ 750/mm^3 (transfusion independent)
* Platelet count* ≥ 50,000/mm^3 (20,000/mm^3 if stem cells are available and platelet transfusion independent)
* Hemoglobin* ≥ 10 g/dL (transfusion allowed)
* No dyspnea at rest
* No exercise intolerance
* No oxygen requirement
* No clinically significant cardiac dysfunction
* No disease of any major organ system that would preclude study compliance
* No active infection that meets grade 3 or 4 toxicity criteria NOTE: *Patients with granulocytopenia and/or thrombocytopenia due to tumor metastases to the bone marrow may be eligible at the discretion of the principal investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 2 weeks since prior antitumor therapy
* At least 3 months since prior radiotherapy to any of the following fields:

  * Craniospinal
  * Total abdominal
  * Whole lung
  * Total body
* At least 1 day since prior cytokine therapy (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], interleukin-6, or epoetin alfa)
* Prior iodine I 131 metaiodobenzylguanidine allowed provided it was given more than 6 months ago AND patient has adequate hematopoietic stem cells available
* No concurrent hemodialysis

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2005-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Ability of iodine I 131 metaiodobenzylguanidine to provide palliative therapy
Acute and late toxicities

SECONDARY OUTCOMES:
Disease and symptom responses

CONTACTS AND LOCATIONS:
Overall Officials: Katherine K. Matthay, MD, Study Chair — University of California, San Francisco; John M. Maris, MD — Children's Hospital of Philadelphia; Robert Goldsby, MD — University of California, San Francisco
Locations (3):
- United States (3):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Matthay KK, Yanik G, Messina J, Quach A, Huberty J, Cheng SC, Veatch J, Goldsby R, Brophy P, Kersun LS, Hawkins RA, Maris JM. Phase II study on the effect of disease sites, age, and prior therapy on response to iodine-131-metaiodobenzylguanidine therapy in refractory neuroblastoma. J Clin Oncol. 2007 Mar 20;25(9):1054-60. doi: 10.1200/JCO.2006.09.3484. PMID 17369569